CLINICAL TRIAL: NCT00245830
Title: Ischemic Preconditioning of Liver in Cadaver Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0120010348
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Liver Cirrhosis; Liver Disease
Keywords: Ischemia/reperfusion of the liver; Ischemic Preconditioning; Cadaver organ donor
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Ischemia | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Hepatic Ischemic Preconditioning (No Intervention): donor will act as a sham control.
- Hepatic Ischemic Preconditioning (Experimental): blood flow to the liver will be cut off by hilar clamping for ten minutes followed by release of the clamp prior to removal of the liver from the donor.
  Interventions: Procedure: Ischemic Preconditioning

INTERVENTIONS:
Procedure: Ischemic Preconditioning — Experimental: Hepatic Ischemic Preconditioning blood flow to the liver will be cut off by hilar clamping for ten minutes followed by release of the clamp prior to removal of the liver from the donor.
  Arms: Hepatic Ischemic Preconditioning

SUMMARY:
The long-term goals of this proposal are to develop clinical protocols of donor preconditioning to improve liver graft function and ameliorate complications of poor graft function after liver transplantation. Achievement of these objectives would improve liver recipient outcomes, increase utilization of livers and alleviate the current critical shortage of livers for transplantation. More stringent liver donor selection intended to decrease the complications of poor graft function conflicts directly with efforts to maximize the use of donor livers. Ischemic preconditioning (IPC) of liver attenuates hepatic ischemia reperfusion injury (IRI) in animals. Preliminary data show hepatic IPC effectively decreases IRI following hepatic resection in humans.

The specific aims of this project are: AIM 1: To test the hypothesis that 10 minutes of hepatic ischemic preconditioning in deceased donors would improve liver graft function and decrease injury in the early post transplant period. AIM 2: To test the hypothesis that ischemic preconditioning of deceased donor livers would decrease systemic inflammatory response in liver recipients in the early post transplant period. AIM 3: To examine whether ischemic preconditioning of deceased donor livers decreases early post transplant pulmonary edema and acute rejection and shortens hospital stay.

DETAILED DESCRIPTION:
Specific Aims

1. To test the hypothesis that 10 minutes of hepatic ischemic preconditioning in deceased donors would improve liver graft function and decrease injury in the early post transplant period.

   To accomplish this aim, we will compare International Normalized Ratios of prothrombin time (INR/PT) and serum aspartate (AST) and alanine aminotransferase (ALT) and total bilirubin (TB) levels immediately post transplant and on day 1, 3, 7, 14 and 30 and injury score of reperfusion liver biopsies in recipients of livers from IPC and No IPC donors.
2. To test the hypothesis that ischemic preconditioning of deceased donor livers would decrease the systemic inflammatory response in liver recipients in the early post transplant period.

   To accomplish this aim, we will compare plasma levels of cytokines tumor necrosis factor-alpha (TNF-alpha), interleukins-6, 8 and 10 (IL-6, 8 and 10) and soluble L-selectin, expression levels of adhesion molecules (CD11beta/CD18 and L-selectin) and oxidative burst of neutrophils, platelet P-selectin and platelet-neutrophil complexes (PNC) in the peripheral blood 3, 12, 24 and 48 hours following reperfusion in recipients of livers from IPC and No IPC donors.
3. To examine whether ischemic preconditioning of deceased donor livers decreases early post transplant pulmonary edema and acute rejection and shortens hospital stay.

To accomplish this aim, we will compare interstitial and alveolar edema in chest radiographs done after transplant and on post operative days 1, 2 and 3; biopsy confirmed acute rejection within 30 days post transplant, and number of days to discharge after transplantation in recipients of livers from IPC and No IPC donors.

Research Design A prospective, randomized, and single masked (liver recipients) study will be conducted in one liver transplant center over a period of two years. Deceased liver donors will be randomized in equal proportions to one of two organ recovery procedures: 1). IPC or 2). No IPC. Allocation will be stratified by age < 50 or age >= 50 to facilitate examination of the effects of age on IPC. As the trial will enroll donors over a two-year period, treatment assignments will be balanced over blocks of length 12, 16 and 20, where the length will be selected at random, to control for time varying factors. Recovered livers are transplanted into recipients > 18 years of age. All other aspects of donor management, organ recovery and preservation, recipient selection, graft implantation and post transplant management including immunosuppression will be according to standard practice.

II. Research Methods

1. Liver Recovery and IPC: Donors are positioned supine, mechanically ventilated and administered 100% oxygen and a muscle relaxant. The abdomen and chest are opened in the midline. Briefly, round and falciform ligaments are divided and the gallbladder is incised and irrigated. The gastroduodenal artery is ligated and junction of splenic and superior mesenteric veins or, when pancreas is procured, the inferior mesenteric vein is prepared for canulation. The supraceliac aorta is exposed just below the diaphragm. The infrarenal abdominal aorta is isolated for canulation. No mobilization of the kidneys is performed before organ perfusion. Thoracic organs are mobilized either simultaneously or before mobilization of abdominal organs. Five hundred units/kg of heparin is given intravenously and ascending thoracic and infrarenal abdominal aorta are canulated. Another canula is inserted either into splenic vein or inferior mesenteric vein. The supraceliac abdominal aorta is clamped and the inferior vena cava is vented in the pericardium. UW solution (40C) is infused into abdominal aorta and portal vein (2 liters each). The abdominal cavity is packed with ice slush. Following completion of organ perfusion heart, lungs, liver and pancreas and kidneys are removed in sequence. Livers are placed in plastic bags containing a liter of UW solution (40C) and packed in ice until the time of transplantation.

   Ischemic preconditioning is performed soon after opening the abdomen by clamping the hepatic hilum with a vascular clamp for five minutes, which is repeated again after five minutes of reperfusion. During IPC the peritoneal cavity is inspected for bleeding, congestion and edema of the pancreas and small intestine.
2. Graft Implantation: Recipient hepatectomy is done in a standard manner with caval preservation and without utilization of venovenous bypass. The liver graft is implanted in a piggyback manner88. The allograft is reperfused after completion of the suprahepatic caval and portal vein anastomoses. The graft is flushed with approximately 300 ml of recipient blood, which is vented via the donor's infrahepatic vena cava, after which this structure is ligated. Arterial and bile duct anastomoses are completed after graft reperfusion.
3. Liver Biopsy and Reperfusion Injury: A wedge and a needle biopsy of the right lobe is performed immediately upon opening the donor's abdomen and before IPC. Another wedge and needle biopsy is done 90 min after recipient reperfusion. Liver biopsy after transplantation is performed only when clinically indicated. Formalin fixed specimens are embedded in paraffin, sectioned five microns thin and stained with hematoxylin and eosin. The amount of fat in donor biopsies is graded semi-quantitatively as follows89; No fat = grade 0, 1-15% = grade I, 16-30% = grade II, 31-45% = grade III, > 45% = grade IV. Reperfusion injury is graded (0-10 in increasing severity) by examining 30 high power fields (600x) of each post perfusion biopsy. Apoptotic cells are enumerated and hepatocyte swelling, zone 3 hemorrhage and necrosis are assigned a semi-quantitative score90. The reperfusion scores in the proposed study are expected to range 0.5 to 5 based on our previous work36. The pathologist is masked regarding the group assignment of all biopsies.
4. Immunosuppression and Acute Rejection: All patients receive tacrolimus and steroids for immunosuppression. In patients with hepatorenal syndrome tacrolimus use is delayed for several days and may be used at a much lower dose than the standard use. Pharmacological immunosuppression will be quantified by determining the mean dose of steroid per day, the mean of the weekly median tacrolimus level for the first five weeks and the proportion of recipients in each group that might receive other agents such as mycophenolate and IL-2 receptor antibody. Immunosuppresion caused by recipient's liver failure will be assessed by their model for end stage liver disease (MELD) score at the time of transplantation. Following transplantation liver biopsies are performed only when clinically indicated. Acute cellular rejection is diagnosed when at least two of the three following criteria are present: portal mononulclear infiltration, bile duct inflammation/damage and subendothelial inflammation of the portal venules and/or terminal hepatic venules. Severity of the rejection is graded based on the rejection activity index as follows: 0-2 = no rejection, 3 = borderline, 4-5 = mild, 6-7 = moderate and 8-9 = severe91. Mild rejection is treated initially with escalation of prograf dose alone or in combination with steroids. Steroid resistant rejection, upon confirmation with a biopsy is treated with muromonab (OKT3).
5. Plasma TNF-alpha, IL-6 and 8, and soluble L-selectin: Plasma is separated from systemic venous blood taken 3, 12, 24, 48 hours after reperfusion from recipients of livers with and without IPC and samples are stored at -700C. TNF-alpha, IL-6 and IL-8 and soluble L-selectin levels are quantitated with commercially available enzyme-linked immunosorbent assay kits (R & D Systems, Minneapolis, MN) in duplicates. The assays are performed according to manufacturer's instructions.
6. Neutrophil CD11beta/CD18 and L-selectin, Platelet P-selectin and Platelet-Neutrophil Complexes and Oxidative burst of Neutrophils in peripheral blood: Systemic venous blood is collected into heparinized (10 U/ml) syringes 3, 12, 24 and 48 hours after reperfusion from recipients of livers with and without IPC. Fifty microL of blood are added to saturating concentrations of fluorescein isothiocyante (FITC), or phycoerythrin (PE) conjugated monoclonal antibodies (Dako Corp, Carpenteria, CA) to CD 11beta/CD18, CD 62 L (L-selectin), CD 42 (platelet von Willebrand factor receptor), and CD 62P (P-selectin). Following 10 min of incubation at room temperature, red cells are lysed by the addition of 200 microL of FACSlyse (Becton Dickinson, Franklin Lakes, NJ). After 10 min of incubation 250 microL of 0.2% formaldehyde in PBS is added. Samples are analyzed in a FasCalibur flow cytometry (Becton Dickinson, Fair Lakes, NJ). Fluorescence of FITC is measured at 515 nm and PE at 580 nm. Neutrophils are distinguished by their readily identifiable characteristics on forward and side-scatter plot. A minimum of 5000 neutrophil events are counted. Events staining positive for both CD 11beta and CD 42 are considered to be PNC as described by Peters et al72. To minimize the risk of identifying individual platelets and neutrophils as PNC flow rate is adjusted to result in < 4500 events/sec. Results are considered positive if the fluorescence intensity exceeds 98% of isotype matched control antibodies. Results are expressed as median fluorescence intensity (MFI). Oxidative burst is measured by utilization of oxidation of dihydrorhodamine to florescent rhodamine by neutrophil generated reactive oxygen species as described by Vowells et al92. Briefly, 300 microL of heparinized whole blood is added to 4 ml of red cell lysis buffer (370C). After five minutes of incubation the pellet is resuspended in HBSS containing 5% fetal calf serum. 1.8 microL of DHR in DMSO is added and incubated at room temperature for 10 min followed by flow cytometric analysis. Stimulation with PMA (1microg/ml) is used as a positive control.
7. Pulmonary Edema: Chest radiographs are performed in an antero-posterior projection with the patient in semi-erect position upon completion of the transplant and on postoperative days 1, 2 and 3. Pulmonary edema is assessed by the presence or absence of interstitial edema and alveolar edema as per accepted criteria93. The radiologist is masked regarding group assignment of subjects.

ELIGIBILITY:
Inclusion Criteria:

- Deceased donor livers allocated to adult (> 18 years of age) recipients at the research site.

Exclusion Criteria:

1. Deceased donor livers allocated to recipients at centers other than the research site.
2. Deceased donor livers allocated to recipients < 18 years of age at the research site.
3. Non-heart beating donors
4. Deceased liver and small intestine donors
5. Live liver donors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Changes in INR/PT and serum AST, ALT and TB levels | Values immediately post-transplantation and on days 1 - 3 and days 7, 14 and 30 post-transplantation

SECONDARY OUTCOMES:
Plasma levels of cytokines | Blood samples are collected at pre-incision of abdomen, cross-clamp of abdominal aorta; 3 hour postreprofusion and post-transplant day one in the recipient
Interstitial and alveolar edema in chest radiographs | days 1 - 3 post transplant
Length of Hospital stay | number of days from Liver transplant to hospital discharge on average 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Baburao Koneru, M.D., Principal Investigator — UMDNJ-New Jersey Medical School
Locations (1):
- University Hospital, Newark, New Jersey, United States

REFERENCES:
- [Background] Koneru B, Fisher A, He Y, Klein KM, Skurnick J, Wilson DJ, de la Torre AN, Merchant A, Arora R, Samanta AK. Ischemic preconditioning in deceased donor liver transplantation: a prospective randomized clinical trial of safety and efficacy. Liver Transpl. 2005 Feb;11(2):196-202. doi: 10.1002/lt.20315. PMID 15666380
- [Background] Raza A, Dikdan G, Desai KK, Shareef A, Fernandes H, Aris V, de la Torre AN, Wilson D, Fisher A, Soteropoulos P, Koneru B. Global gene expression profiles of ischemic preconditioning in deceased donor liver transplantation. Liver Transpl. 2010 May;16(5):588-99. doi: 10.1002/lt.22049. PMID 20440768
- [Background] Desai KK, Dikdan GS, Shareef A, Koneru B. Ischemic preconditioning of the liver: a few perspectives from the bench to bedside translation. Liver Transpl. 2008 Nov;14(11):1569-77. doi: 10.1002/lt.21630. PMID 18975290
- [Result] Koneru B, Shareef A, Dikdan G, Desai K, Klein KM, Peng B, Wachsberg RH, de la Torre AN, Debroy M, Fisher A, Wilson DJ, Samanta AK. The ischemic preconditioning paradox in deceased donor liver transplantation-evidence from a prospective randomized single blind clinical trial. Am J Transplant. 2007 Dec;7(12):2788-96. doi: 10.1111/j.1600-6143.2007.02009.x. Epub 2007 Oct 19. PMID 17949458